CLINICAL TRIAL: NCT07232901
Title: Implementing Family Participation Training in Tertiary Hospital Care in Bangladesh: a Stepped-wedge Realist Trial
Brief Title: Implementing Family Participation Training in Tertiary Hospital Care in Bangladesh
Acronym: FAMCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele van Vugt (Other)
Collaborators: Chittagong Medical College and Hospital (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Asian University for Women (Unknown); Noora Health (Unknown); Mixit (Unknown); Amsterdam UMC (Other)
Responsible Party: Sponsor-Investigator, Michele van Vugt, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: FAMCARE
Record Dates: First submitted 2025-09-02; First posted 2025-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Family Participation in Hospital Care; Hospital Medicine; Training Family Caregivers
Keywords: Caregiver; Family; Hospital; Nursing; Co-creation; Stepped-wedge; Realist Evaluation; Training; Implementation; Participation

STUDY DESIGN:
Intervention Model Description: Stepped-wedge trial
Masking Description: Unable to mask a training intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Control: Hospital care as usual.
- Family Caregiver Training (Experimental): Intervention: Family Caregiver Training in hospital.
  Interventions: Behavioral: Family Caregiver Training

INTERVENTIONS:
Behavioral: Family Caregiver Training — This study will test a family participation training intervention. Family caregivers will receive training on participating in hospital care while nurses and doctors receive training to train family caregivers. The family caregiver training sessions will be delivered during the intervention period in three wards to all family caregivers willing to attend the training session. The intervention has been co-created and piloted with patients, family caregivers, health workers, and hospital administrators. The content of the training will include an introduction to the hospital environment, basic care tasks, warning sign detection, oral medication administration, caregiver handover, and discharge preparedness. The content of the family caregiver training will be bundled in a visual poster. These posters will be hung on the walls across the medicine wards at the patients' bedsides.
  Arms: Family Caregiver Training

SUMMARY:
The goal of this trial is to evaluate whether a family participation training intervention can reduce caregiver strain and health worker workload, and improve patient outcomes and collaboration in the medicine wards of Chittagong Medical College Hospital (CMCH).

General objectives:

* To assess the effect of a family participation training intervention on the medicine wards of CMCH. (Stepped-wedge)
* To examine how, for whom and under what circumstances a family participation training intervention works. (Realist evaluation)

Specific objectives:

* To examine the implementation of a family participation training intervention.
* To investigate the acceptability and feasibility of a family participation training intervention.

The study will use a step-by-step roll-out, introducing training at different times in three wards, to see if it improves care compared to usual practice.

Study participants will include adult patients, their family caregivers, nurses, doctors, ward assistants, and hospital administrators. Health workers will be trained to deliver sessions to family caregivers of hospitalised patients on hospital introduction, basic care tasks, warning sign detection, oral medication administration, caregiver handover, and discharge preparedness.

DETAILED DESCRIPTION:
Background:

In many resource-limited settings, understaffed hospitals rely on the families of patients to provide care during admission. Family participation in hospital care may include washing, toileting, feeding, administering medication, and detecting warning signs. Family participation in hospital care is commonplace at Chittagong Medical College Hospital (CMCH) and other hospitals in Bangladesh. These care tasks are often performed informally, untrained, and unsupported, resulting in a high mental and physical burden of care for family caregivers, unknown effects on patient outcomes and potentially an even higher workload for health workers. This study proposes to implement and evaluate a family participation training intervention in the general medicine wards of CMCH. Building on prior preparatory research, the intervention aims to reduce family caregiver strain, lower health workers' workloads, enhance patient outcomes and improve collaboration between family caregivers and health workers.

Objective The primary objectives of the study are to assess the effect of a family participation training intervention on the medicine wards of CMCH and to examine how, for whom and under what circumstances a family participation training intervention works.

Methods The study employs a stepped-wedge realist trial over six months in the CMCH medicine wards (13, 14, and 16). It involves adult patients, family caregivers, health workers (nurses, doctors, and ward assistants), and hospital administrators. Family caregivers will receive training to support their participation in hospital care, while nurses and doctors will be trained to deliver these sessions. The training will include an introduction to the hospital, basic hospital care, oral medication administration, detection of warning signs, handover between family caregivers, and discharge preparation. The primary outcomes are reduced family caregiver strain and lower health worker workload. Patient-family caregiver dyads will be followed daily for up to five days during admission and one call after discharge. Health workers will be followed throughout the study period. In addition, ward-level, implementation, feasibility, and acceptability outcomes will be collected. Some patients, family caregivers, health workers, and hospital administrators will be included in realist interviews or focus group discussions. The analysis will integrate mixed-effects modelling with a realist evaluation approach.

Discussion This study will add a foundational piece of research to the family participation field, in resource-limited and -rich settings. It builds on the shared journey of this growing international research collaboration. No such previous research has been performed. It will be the first to test a co-created family participation training intervention in hospital care. In addition, it suggests new research methods by integrating a stepped-wedge design with a realist evaluation.

ELIGIBILITY:
Inclusion Criteria:

All study parts

Population

* Patient: admitted to one of the three medicine ward
* Family caregiver: caregiver providing care for a patient on one of the three medicine wards
* Health worker: nurse, doctor or ward assistant working on one of the three medicine wards
* Hospital administrator: professors or administrators responsible for or directly involved in policymaking or have operational oversight on one of the three medicine wards

Adult

- Age: ≥18 years

Data collection specific Patient and family caregiver data collection - Patient & family caregiver dyad: admitted for ≤24 hours on the medicine wards

Health worker data collection

- Employment: working on one of the medicine wards for at least one week

Interviews, focus group discussions and observations

* Patient: admitted ≥24 hours on the medicine wards
* Family caregiver: caring for the patient ≥24 hours on the medicine wards

During the intervention period

* Patient: family caregiver of the patient has received the training
* Family caregiver: has received the training

Exclusion Criteria:

All

Language - Unable to speak Bengali, Chittagonian or English

Consent

* No consent given
* Unable to give consent
* Duplicates: Previously enrolled in the study

Data collection specific Patient and family caregiver data collection

- Patient: Planned discharge ≤24 hours of admission to the medicine ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2025-08-09 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Family Caregiver: Strain | During 5 day hospital follow-up
  Measured with Care-related Quality of Life (CarerQOL), ranging from 0 (worst care situation) to 100 (best care situation)
Health Worker: Workload | Assessed from inclusion till study end for at least once per study period across four periods, spanning five months in total
  Nasa Task Load Index, ranging from 0 (low workload) to 10 (high workload)
Refined Programme Theories from the Realist Evaluation | Continuous refinement from start of the intervention till end of the study, spanning four months in total
  The refined programme theories will be developed through iterative analysis of qualitative and quantitative data, outlining what works in the intervention, for whom, and under what circumstances.

SECONDARY OUTCOMES:
Family Caregiver: Workload | During 5 day hospital follow-up
  Nasa Task Load Index, ranging from 0 (low workload) to 10 (high workload)
Family Caregiver: Caregiving Tasks Performed During Hospitalisation | During 5 day hospital follow-up
  Daily collection of which caregiving tasks were performed in the past 24 hours by the main family caregiver, other family caregivers and the patient themselves.
Family Caregiver: Readiness for Discharge | During 5 day hospital follow-up
  The caregiver is asked daily how ready they would be to provide care at home if their relative would be discharged today.
Family Caregiver: Satisfaction with Hospital Care | During 5 day hospital follow-up and at 14 day call
  Adapted and shortened HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) Survey, measured on a four and ten point scale
Health Worker: Families' Importance in Nursing Care | Assessed from inclusion till study end for at least once per study period across four periods, spanning five months in total
  Using the Families' Importance in Nursing Care - Nurses' Attitudes (FINC-NA), measured on a five point scale
Health Worker: Interruptions | Assessed from inclusion till study end for at least once per study period across four periods, spanning five months in total
  Health workers are asked about their perceived increase or decrease in interruptions during work by family caregivers

OTHER OUTCOMES:
Patient: Satisfaction with Hospital Care | During 5 day hospital follow-up
  Adapted and shortened HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) Survey, measured on a four and ten point scale
Patient: Anxiety and Depression | During 5 day hospital follow-up
  Patient Health Questionnaire-4 (PHQ-4), measured on a four point scale
Patient: Readiness for Discharge | During 5 day hospital follow-up
  Patient Readiness for Discharge Scale, measured from 0 (worst) to 10 (best) readiness
Patient: Medication Adherence | During 5 day hospital follow-up
  Pill counts
Patient: Hospitalisation Outcomes | During 5 day hospital follow-up and 14 day call
  Outcome of hospital admission: discharged home alive, left against medical advice, in another hospital, died in hospital, discharged home to die, in ICU, in another ward, still in the medicine ward, lost to follow-up.
Implementation: Reach | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Training logs recording all family caregivers and patients trained
Implementation: Adoption | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Uptake of the intervention by health workers and the ward.
Implementation: Fidelity | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Fidelity sheets of the training sessions
Implementation: Adaptions | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Modifications made during implementation of the intervention
Implementation: Cost of the Intervention | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Resources required to deliver the intervention
Feasibility & Acceptability | Continuous data collection from the start of the intervention until the end of the study (four months in total).
  Qualitative assessment of integration of the training intervention into the health worker and ward workflow, resource feasibility of the intervention, buy-in from stakeholders and feasibility of the research methods for this intervention type.

CONTACTS AND LOCATIONS:
Overall Officials: Michèle van Vugt, Prof. Dr., Principal Investigator — Amsterdam University Medical Center
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: No